CLINICAL TRIAL: NCT07381582
Title: A Prospective, Open-label, Dose-Escalation, Single-Center Study to Evaluate the Safety, Biodistribution/Dosimetry and Preliminary Efficacy of 161Tb-LNC1011 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Safety, Tolerability and Preliminary Efficacy of 161Tb-LNC1011 (PSMA Radioligand) in Patients With Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Acronym: 161Tb-LNC1011
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Mianyang Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-MCH-161Tb-LNC1011
Record Dates: First submitted 2025-11-23; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Terbium-161; PSMA; Radionuclide therapy; Metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Intravenous administration; planned dose levels: 50, 80, 130, 200 mCi (±10%); cycle interval q6 weeks; up to 1 cycle at 50 mCi and up to 4 cycles at later dose levels as permitted by safety and disease status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-Escalation Cohort (3+3): 161Tb-LNC1011 (Experimental): Single-group, open-label, sequential dose escalation of 161Tb-LNC1011 (IV). Planned dose levels: 50, 80, 130, 200 mCi (±10%). At 50 mCi: 1 cycle; higher levels: up to 4 cycles every 6 weeks, contingent on safety and disease status. DLT window: 6 weeks post-dose; MTD per standard 3+3 rules (≥2/6 DLTs defines exceeding dose). Retreatment requires hematologic recovery to CTCAE ≤ Grade 1 or baseline. Post-dose SPECT/CT at ~30 min, 2 h, 8 h, 24 h, Day 2, Day 7 for dosimetry; disease assessments with 68Ga-PSMA-11 PET/CT and labs per schedule.
  Interventions: Drug: 161Tb-LNC1011

INTERVENTIONS:
Drug: 161Tb-LNC1011 — Intravenous administration; planned dose levels: 50, 80, 130, 200 mCi (±10%); cycle interval q6 weeks; up to 1 cycle at 50 mCi and up to 4 cycles at later dose levels as permitted by safety and disease status.

SUMMARY:
This is a prospective, open-label, single-center, dose-escalation study using a standard 3+3 design to assess the safety, tolerability, biodistribution/dosimetry and preliminary efficacy of the albumin-binding PSMA radioligand 161Tb-LNC1011 in patients with metastatic castration-resistant prostate cancer (mCRPC). Patients will receive intravenous 161Tb-LNC1011 starting at 50 mCi with planned dose-level escalations to 80, 130 and 200 mCi (±10%). Early dose levels (50 mCi) receive 1 cycle; later levels receive up to 4 cycles every 6 weeks based on safety and disease status. Primary endpoints include dose-limiting toxicities (DLTs), adverse events (AEs) graded by CTCAE v5.0, and determination of maximum tolerated dose (MTD). Secondary endpoints include organ/tumor absorbed doses, PSA responses (PSA50/PSA90), disease control, time to PSA progression and radiographic progression-free survival per PCWG3.

DETAILED DESCRIPTION:
Rationale: 161Tb emits β-particles plus abundant low-energy conversion/Auger electrons (very short range, high LET), potentially improving tumoricidal effect-especially for micrometastases-vs 177Lu. LNC1011 is a PSMA ligand with albumin-binding moiety designed to prolong circulation and enhance tumor uptake/retention. Preclinical and early clinical data support feasibility and safety.

Design: 3+3 dose-escalation. Dose levels (activity to be administered IV): 50 mCi (45-55), 80 mCi (72-88), 130 mCi (117-143), 200 mCi (180-220). DLT window: 6 weeks post-dose. If ≥2/6 DLTs, de-escalate; the prior dose is MTD.

Dosing/Cycles: Early dose level (50 mCi) one cycle; later levels up to 4 cycles q6 weeks. Retreatment contingent on hematologic recovery to CTCAE Grade ≤1 or baseline.

Imaging & Dosimetry: Post-dose SPECT/CT at ~30 min, 2 h, 8 h, 24 h, Day 2, Day 7 for time-activity curves and dosimetry. Disease assessments with 68Ga-PSMA-11 PET/CT and labs (PSA, hematology, chemistry) per schedule.

Safety Monitoring: Continuous AE/SAE recording from consent through 28 days post-last dose (or longer if related), DMC oversight (see below).

ELIGIBILITY:
Inclusion Criteria:

* Male, ≥18 years.
* Pathologically confirmed mCRPC per PCWG3.
* 68Ga-PSMA-11 PET/CT positive.
* Prior exposure to at least one novel androgen-axis drug (e.g., enzalutamide and/or abiraterone) or at least one taxane regimen, or intolerance/refusal to taxane chemotherapy.
* ECOG 0-2; life expectancy ≥6 months.
* Adequate organ function: ALT/AST ≤3× ULN; BUN/Cr ≤1.5× ULN; WBC ≥3.5×10^9/L; PLT ≥100×10^9/L; Hb ≥90 g/L.
* Signed informed consent and willingness to comply with study procedures.

Exclusion Criteria:

* Major trauma/surgery within 4 weeks prior to study treatment.
* Active severe systemic or localized infection or other serious comorbidity.
* Immunodeficiency or recent use of immunosuppressants/immunoenhancers, recent vaccines.
* Autoimmune diseases (e.g., rheumatoid arthritis) requiring active management.
* Uncontrolled arrhythmias (incl. Afib), heart failure NYHA > II, uncontrolled hypertension.
* Known allergy to components of investigational product.
* Positive syphilis, HBV/HCV/HIV.
* Inadequate contraception in patients of reproductive potential.
* Psychiatric illness compromising compliance.
* Unable to undergo SPECT/CT or to retain urine for 30 minutes.
* Any condition deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | First 6 weeks after each initial dose at a given dose level
  Proportion of participants with DLTs per CTCAE v5.0 during the DLT window.
Maximum Tolerated Dose (MTD) | At completion of dose escalation (approximately 12-18 months after study start)
  Highest dose level at which ≤1/6 participants experience a DLT.
Treatment-Emergent Adverse Events (TEAEs) | From first dose through 28 days after last dose (extended if related)
  Number and grade of AEs/SAEs per CTCAE v5.0.

SECONDARY OUTCOMES:
Organ and Tumor Absorbed Doses (Dosimetry) | Within first cycle (Day 0 to Day 7 imaging)
  Absorbed doses to kidneys, salivary glands, tumor lesions, etc., derived from serial SPECT/CT.
PSA50 and PSA90 Response Rates | Every 6 weeks during treatment and at end of treatment (up to approximately 24 weeks)
  Proportion achieving ≥50% and ≥90% PSA decline from baseline, confirmed per PCWG3.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Mianyang Central Hospital, Mianyang, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided